CLINICAL TRIAL: NCT02624453
Title: Implementation and Evaluation of a Screening Strategy to Reduce Morbidity and Mortality Due to Cryptoccocal Meningo-encephalitis in ART Naive AIDS Patients With <100 CD4 Count at the Day Hospital of the Yaounde Central Hospital, Cameroon
Brief Title: Pre-Antiretroviral Therapy (ART) Cryptococcal Antigen Screening in AIDS
Acronym: PreCASA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Yaounde Central Hospital (Other Government); St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: ANRS 12312 PreCASA
Record Dates: First submitted 2015-12-04; First posted 2015-12-08 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Cryptococcal Meningitis
Keywords: cryptococcus; IMMY LFA; meningitis; antigen
MeSH Terms: conditions — Meningitis, Cryptococcal; Meningitis | interventions — Fluconazole; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMMY LFA positive patients (Experimental): HIV positive patients who will be positive for cryptococcal antigen (by the IMMY LFA test) would be consented for lumbar puncture in search of cryptococcal meningitis (CM). If CM is not confirmed, they would be prescribed pre-emptive fluconazole based therapy at 800mg/day for two weeks (placed on antiretroviral therapy two weeks after screening for cryptococcal antigen), then 400mg/day for 8 weeks and thereafter 200mg/day until CD4 counts increases beyond 200cells/ml. (CM confirmed cases will be referred to the ACTA trial ISRCTN45035509)
  Interventions: Drug: Fluconazole; Drug: Antiretroviral therapy
- IMMY LFA negative patients (Active Comparator): HIV positive patient who will be negative for cryptococcal antigen (by the IMMY LFA test) would not be consented for lumbar puncture, will be placed immediately on antiretroviral therapy immediately after screening for cryptococcal antigen and would not be placed on fluconazole pre-emptive therapy.
  Interventions: Drug: Antiretroviral therapy

INTERVENTIONS:
Drug: Fluconazole — Pre-emptive fluconazole therapy at 800mg/day for two weeks, then 400mg/day for eight weeks, and then 200mg/day thereafter till CD4 count goes beyond 200cells/ml
  Other Names: cryptococcal antigen positive patients
  Arms: IMMY LFA positive patients
Drug: Antiretroviral therapy — First line anti-retroviral therapy according to Cameroon national guidelines for the management of HIV/AIDS
  Other Names: cryptococcal antigen negative patients

SUMMARY:
The aim of the study is to evaluate systematic pre-antiretroviral cryptococcal antigen screening and pre-emptive fluconazole therapy in antigen positive patients, as a strategy to reduce morbidity and mortality due to AIDS associated cryptococcal meningitis in patients starting antiretroviral therapy at <100 CD4 in Cameroon.

DETAILED DESCRIPTION:
Cryptococcal meningitis (CM) is a leading cause of death in AIDS patients in much of the developing world, responsible for up to 500,000 deaths each year in sub-Saharan Africa alone. Introduction of antiretroviral therapy (ART) has reduced the number of cases of cryptococcal meningitis in the developed world. Unfortunately, in many low resource settings, patients continue to present late to ART treatment programs with advanced immunosuppression, and many die of HIV-related illness in the weeks just prior to, and months following, initiation of ART. Cryptococcal meningitis causes many of these deaths, and is also a heavy burden on healthcare facilities. Treatment of the disease remains inadequate, with an acute mortality of between 20 and 50%, even with the best current treatment.

Many of these cases of cryptococcal meningitis may be preventable. Recent research has shown that routine screening for sub-clinical infection, using a simple test (cryptococcal antigen or CRAG) in patients presenting to ART programmes, can identify which patients are at risk of developing cryptococcal meningitis. Once identified, these patients could then be given safe oral "pre-emptive" treatment to prevent them developing a severe form of the disease. This strategy has many advantages over the alternative preventative measure, called generalised primary prophylaxis, which involves giving all profoundly immune depressed HIV-infected patients preventative treatment. Using a primary prophylaxis strategy, large numbers of patients are given medication, many of whom don't need it, and there are problems of cost and development of drug resistance and drug interactions. In a targeted strategy, only patients who benefit most from the treatment will be given medication.

The investigators propose to study the feasibility and effectiveness of CRAG screening and targeted pre-emptive treatment in patients entering ART treatment programmes in Yaoundé, Cameroon using a newly approved, easier to use, lateral flow format dipstick test (LFA). In the planned study, 400 patients will be screened using the CRAG test prior to starting ART. Patients with a positive cryptococcal antigen will be consented for a lumbar puncture (LP) for cerebrospinal fluid (CSF) analysis, and, if found to have cryptococcal meningitis, and eligible, they will be randomised and included in the complementary clinical trial "Advancing Cryptococcal Treatment in Africa" (ACTA) [ISRCTN45035509, ANRS12275] and treated according to the study protocol. Positive cryptococcal antigen patients with no evidence of neurological disease following lumbar puncture, or who decline a diagnostic LP will receive a tapering course of fluconazole. Cryptococcal antigen negative patients will not receive any additional antifungal therapy. All CRAG screened patients will be started on standard ART 2 to 4 weeks after screening and followed for up to 1 year, depending on antigen status, to determine whether any patients go on to develop clinical cryptococcal meningitis.

General objective

- To implement and evaluate systematic cryptococcal antigen screening as a strategy to reduce cryptococcal meningoencephalitis morbidity and mortality among HIV-infected patients initiating antiretroviral therapy at less than 100 CD4 cell counts at the Day Hospital of the Yaoundé Central Hospital in Cameroon

Specific objectives

* To determine the prevalence of cryptococcal antigenaemia and/or antigenuria among HIV-infected patients presenting with less than 100 CD4 cell count
* To determine the prevalence of laboratory confirmed cryptococcal meningoencephalitis among patients found to be CRAG positive
* To determine the incidence of newly diagnosed, and relapsing, laboratory confirmed cryptococcal meningitis in the first year after starting ART in all screened patients.
* To determine mortality within the first year of ART among patients screened for CRAG

Study design and number of patients A prospective cohort study of 400 ART naive patients presenting at entry of ART programme with less than 100 CD4 cell count/ml will be screened for CRAG using LFA in serum and urine and followed up for one year.

Study interventions Main intervention of the study will be cryptococcal antigen (CRAG) screening. All eligible patients will be screened at baseline using an LFA, a point of care (POC) dipstick test, on serum and/or plasma, and urine. Aliquots will be saved for later titering of CRAG positive samples. All subsequent treatments and patient management will be according to local guidelines and/or internationally accepted best practice standards.

Subsequent management Cryptococcal antigen negative participants: All CRAG negative participants will commence ART once counselling and pre-ART work-up are complete within an estimated time of 2 weeks in accordance with current Cameroon National AIDS control programme guidelines. There will be no further interventions. The participant will be seen at the outpatient clinic on the 2nd and 4th weeks following screening, then routinely according to the day hospital roster, and finally, every three months up to one year after the date of screening.

Cryptococcal antigen positive participants: All CRAG positive participants will have a careful symptom screen (headache/altered mental status), and will be asked to consent for an LP for CSF analysis: If cryptococcal meningitis is diagnosed by Indian ink and/or culture, and the patients is eligible, the patient may be included in the clinical trial "Advancing Cryptococcal Treatment in Africa" (ACTA) and treated according to ACTA protocol. If a patient is ineligible, or declines to be included in the ACTA trial, they will be treated with short course amphotericin B (one week) combined with oral fluconazole 800mg/day for two weeks, then 8 weeks of fluconazole 40mg/day and 200mg/day thereafter.

If LP is negative for cryptococcal meningitis (or LP refused), patients will receive Fluconazole 800 mg/day for 2 weeks then 400 mg/day for 8 weeks then 200 mg/day (based on current best practice).

Patients will commence ART (efavirenz based) 2-4 weeks after starting antifungal therapy, in accordance with current Cameroon National AIDS control programme guidelines. Follow-up will be for one year. Patients will be seen at the outpatient clinic every two weeks for the first ten weeks, then at three month intervals. During the outpatient visits, in case of any opportunistic infection occurrence, they will be managed according to local current practice of the Day Hospital. Women of child-bearing age will be proposed contraception (preferably barrier methods) during the period of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18years
* HIV 1 and 2 infected but naïve to ART
* CD4 cell count less than 100 cells/ml
* No documented past history of cryptococcal meningoencephalitis
* Acceptance to participate in the study
* Ambulatory/out patients.

Exclusion Criteria:

* Patients on ART
* Pregnant patients
* Patients with other severe AIDS-associated opportunistic infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2015-07; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cryptococcal antigenaemia and antigenuria | at inclusion
  Prevalence of cryptococcal antigenaemia and antigenuria in HIV patients with CD4 ≤ 100 cells/µL at the Day Hospital of the Yaoundé Central Hospital

SECONDARY OUTCOMES:
Baseline prevalence of laboratory confirmed Cryptococcal Meningitis | at inclusion
  Baseline prevalence of laboratory confirmed Cryptococcal Meningitis among patients screened positive for Cryptococcal antigen

OTHER OUTCOMES:
Incidence of laboratory confirmed cryptococcal meningitis in the first year | first year of antiretroviral therapy initial
  Incidence of laboratory confirmed cryptococcal meningitis in patients screen cryptococcal antigen positive in the first year of anti-retroviral therapy
Incidence of newly diagnosed and relapsing in all patients in the first year | first year of antiretroviral therapy initiation
  Incidence of newly diagnosed and relapsing, laboratory confirmed, cryptococcal meningitis in the first year after starting ART in patients screened for cryptococcal antigen.
Incidence of mortality within the first year | first year of antiretroviral therapy initiation
  Incidence of mortality within the first year of antiretroviral therapy among cryptococcal antigen screened patients

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lortholary, MD, PhD, Principal Investigator — Hôpital Universitaire Necker-Enfants Malades, Molecular Mycology Unit, Institut Pasteur of Paris, and Paris Descartes University, Paris, France; Elvis Temfack, MD, MSc, Principal Investigator — Douala General Hospital, Douala, Cameroon and Paris Descartes University, Paris, France; Thomas Harrison, MD, Study Director — Infectious Disease Unit, St George's University of London, London, United Kingdom; Charles Kouanfack, MD, PhD, Study Director — Day Hospital, Yaoundé Central Hospital, Yaoundé, Cameroon
Locations (1):
- Day Hospital of the Yaounde Central Hospital, Yaoundé, Central Region, Cameroon